CLINICAL TRIAL: NCT01514877
Title: Phase II Study of Icotinib Combined With Whole Brain Radiotherapy in Treating Patients With Brain Metastases From Non-Small Cell Lung Cancer
Brief Title: Icotinib Combined With Whole Brain Radiotherapy in Treating Multiple Brain Metastases From Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZhejiangCH-LCBM-1201
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; non-small cell lung cancer; Icotinib
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib plus Whole Brain Radiotherapy (Experimental): Epidermal growth factor receptor (EGFR) tyrosine kinase inhibitors (TKIs), such as gefitinib and erlotinib, have shown efficacy in advanced non-small cell lung cancer (NSCLC) patients with brain metastases (BM). Icotinib is a new first generation EGFR-TKI. We conducted a phase II study to evaluate the efficacy and safety of icotinib in combination with whole brain radiotherapy （WBRT） in Chinese NSCLC patients with BM and investigated the cerebrospinal fluid (CSF)/ plasma concentrations of icotinib.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Patients will receive whole brain radiotherapy therapy 30Gy over 10 fractions and icotinib will be administered at the beginning of whole brain radiotherapy in doses of 125 mg thrice per day until disease progression or undue toxicity.

SUMMARY:
The aim of this study is to explore the efficacy and toxicity of icotinib combined with WBRT in treating patients with multiple brain metastases from NSCLC.

DETAILED DESCRIPTION:
Brain metastases occur in 25-40% of patients with non-small cell lung cancer (NSCLC). It is one of the primary reasons resulting in treatment failure and the death. Whole-brain radiation therapy (WBRT) is the standard approach to the treatment of multiple brain metastases from NSCLC. Regardless of the treatment of brain metastases by WBRT combined with systemic chemotherapy,outcomes of NSCLC with brain metastases are still very poor. Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKIs) can pass through the blood-brain barrier and show promising antitumor activity against brain metastases from NSCLC. Icotinib shows nearly the same effect as gefitinib in advanced NSCLC patients failed with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Cytologic or histological diagnosis of non-small cell lung cancer
* Patients with disease progression after systemic chemotherapy with two-drug combination regimens that includes a platinum agent or patients with EGFR mutation status who have not been treated
* Patients are diagnosed with multiple brain metastases for the first time in 4 weeks
* Diagnosis of brain metastases is made based on Magnetic resonance imaging (MRI).
* Doctors consider the patient will benefit from WBRT
* No prior brain radiotherapy
* ECOG performance status 0-2
* age:18-75 years
* Neutrophil count ≥1.5×10 to the 9th power/L and platelets≥100×10 to the 9th power/L. hemoglobin ≥90 g/L
* Hepatic: total bilirubin less than or equal to 1.5 times upper limit of normal (ULN) Alanine transaminase (ALT) and aspartate transaminase (AST) less than or equal to 2.5 times ULN (or less than or equal to 5 times ULN in case of known liver involvement)
* Renal: Serum Creatinine less than or equal to 1.5 times upper limit of normal (ULN)
* Patients with measurable brain metastases according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study

Exclusion Criteria:

* Prior brain radiation therapy
* Solitary brain metastasis according to Magnetic resonance imaging (MRI)
* Mort than 3 extracranial organs have metastatic lesions
* Prior invasive malignancy (skin basal cell cancer, carcinoma in situ of cervix are permissible).
* pregnant or breast feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
partial response rate of intracranial lesions | 2 years
  Partial response rate of intracranial lesions will be measured.

SECONDARY OUTCOMES:
Progression-free survival | 4 years
  Progression-free survival will be evaluated
overall survival | 4 years
  Overall survival will be evaluated
partial response rate of extracranial lesions | 2 years
  Partial response rate of extracranial lesions will be evaluated
Health-related quality of life | 2 years
  Health-related quality of life will be measured
safety and tolerability | 4 year
  Safety and tolerability of Icotinib and whole brain radiotherapy will be monitored by evaluation of frequency,severity,and duration of treatment-emergent adverse events in all subjects
the relationship between Progression-Free Survival and EGFR mutation status | 4 years
  The relationship between Progression-Free Survival and EGFR mutation status will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yun Fan, MD, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Fan Y, Huang Z, Fang L, Miao L, Gong L, Yu H, Yang H, Lei T, Mao W. A phase II study of icotinib and whole-brain radiotherapy in Chinese patients with brain metastases from non-small cell lung cancer. Cancer Chemother Pharmacol. 2015 Sep;76(3):517-23. doi: 10.1007/s00280-015-2760-5. Epub 2015 Jul 7. PMID 26148750